CLINICAL TRIAL: NCT04834492
Title: At Least 10-Year Results of Cementless Ceramic-On-Ceramic Total Hip Arthroplasty Performed With Transverse Subtrochanteric Osteotomy in Crowe Type 4 Hips.
Brief Title: The Results of Total Hip Arthroplasty in Crowe Type 4 Hips.
Status: Completed | Type: Observational
Sponsor: Private Ortopedia Hospital, Seyhan Adana (Other)
Responsible Party: Principal Investigator, Cagri Ors, Medical Doctor, Private Ortopedia Hospital, Seyhan Adana
Other Study IDs: Crowe type 4
Record Dates: First submitted 2021-04-04; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: The Results of Total Hip Arthroplasty in Crowe Type 4 Dysplastic Hips
Keywords: Developmental dysplasia of the hip, total hip arthroplasty, transverse subtrochanteric shortening osteotomy, ceramic on ceramic, cementless.
MeSH Terms: conditions — Developmental Dysplasia of the Hip | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Total hip arthroplasty — Total hip arthroplasty in Crowe type 4 developmental dysplasia of the hip.

SUMMARY:
Total hip arthroplasty (THA) performed for developmental dysplasia of the hip (DDH) is a technically difficult procedure with a high complication rate, especially in the presence of completely dislocated hips. This study aimed to evaluate the results of at least 10 years of follow-up results of cementless, ceramic-on-ceramic (CoC) total hip arthroplasty performed with transverse subtrochanteric osteotomy in Crowe type 4 hips.

DETAILED DESCRIPTION:
We reviewed retrospectively 67 hips of 50 patients which underwent CoC, cementless THA with transverse subtrochanteric osteotomy between 2008 and 2011. Clinical and radiological data of the hips were examined. Clinical results were evaluated using the Harris Hip Score (HHS) and the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC).

ELIGIBILITY:
Inclusion Criteria:

Crowe type 4 developmental dysplasia of the hip

Exclusion Criteria:

Primary Coxarthrosis

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Crowe type 4 developmental dysplasia of the hip patient
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Clinical results | minimum 10 year follow-up
  Haris Hip Score

CONTACTS AND LOCATIONS:
Locations (1):
- Private Ortopedia Hospital, Adana, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No